CLINICAL TRIAL: NCT00503633
Title: Biomarkers of Insomnia and Fatigue in HIV/AIDS
Brief Title: Biomarkers of Insomnia and Fatigue in HIV/AIDS (Symptoms and Genetics Study)
Acronym: SAG
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Kathryn A. Lee, PhD, University of California, San Francisco
Other Study IDs: SAG
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: HIV Infections
Keywords: sleep disorders; genetics
MeSH Terms: conditions — HIV Infections; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify biological markers, including genes, associated with sleep disturbance and other symptoms among people with HIV.

DETAILED DESCRIPTION:
This study will characterize insomnia subtypes and identify genetic markers and metabolic parameters associated with these subtypes. The results will be useful in later developing interventions to improve sleep, reduce fatigue, and thereby enhance the quality of life of HIV-infected persons.

A cross-sectional sample of 350 subjects will be recruited to describe relationships between biomarkers and insomnia subtypes. The initial assessment will include:

* wearing a wrist actigraph for 72 hours
* providing a fasting blood sample
* measuring blood pressure, height, weight, neck, waist, hip, and thigh
* completing questionnaires
* urine screening

Depending on the results of the initial assessment, approximately 200 subjects will be followed every month by telephone to assess symptoms and every 3 to 6 months with study visits similar to the initial assessment. Findings from this longitudinal part of the study will characterize the development of insomnia, fatigue, and daytime sleepiness over time in patients living with HIV.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Access to a telephone
* Able to read and write English

Exclusion Criteria:

* Current use of illicit drugs
* Currently pregnant or within the previous 3 months
* Working nightshift
* Diagnosis of sleep apnea, narcolepsy, restless legs syndrome, or periodic limb movements, dementia, or psychotic illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with HIV
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2005-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn A Lee, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States